CLINICAL TRIAL: NCT04012801
Title: Evaluation of C13 Breath Test for Upper Gastrointestinal Bleeding in Patients of Acute Myocardial Infarction Who Need Double Antiplatelet After PCI
Brief Title: Evaluation of C13 Breath Test for Upper Gastrointestinal Bleeding in Patients Who Need Double Antiplatelet After PCI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Associate Professor, Chongqing Medical University
Other Study IDs: 2019-09
Record Dates: First submitted 2019-06-22; First posted 2019-07-09 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: C13 breath test — C13 breath test for patients of acute myocardial infarction who need dual- antiplatelet after PCI.

SUMMARY:
Hp infection is closely related to upper gastrointestinal bleeding in patients who need dual-antiplatelet after PCI. Taking anti-Hp treatment has the effect of reducing bleeding risk. Thus, we propose a scientific hypothesis: the C13 breath test may be used to assess the risk of upper gastrointestinal bleeding in patients who need dual- antiplatelet after PCI.

DETAILED DESCRIPTION:
Our study is to retrospectively analyze the clinical data of 1606 patients of acute myocardial infarction who need dual- antiplatelet after PCI.The diagnostic criteria for upper gastrointestinal bleeding is: 1.symptoms: digestive discomfort, such as abdominal pain, nausea, belching, acid reflux, etc.;2.mainly based on endoscopy examination, endoscopic examination showed that the stomach or duodenum showed spotted, linear or diffuse bleeding;3.the fecal examination:melena, tar-like stool, hematemesis, fecal occult blood, etc.The study was divided into two groups according to whether the C13 breath test was performed, and the C13 breath test component was the positive anti-HP treatment group and the non-anti-HP treatment group.And then compare the upper gastrointestinal bleeding rates of the above groups.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of patients with coronary heart disease is based on the diagnostic criteria of ACA/AHA,the diagnostic criteria for upper gastrointestinal bleeding refer to the guidelines for the diagnosis and treatment of acute non-variceal upper gastrointestinal bleeding.
* In the hospital, all patientsI were treated with clopidogrel 300 mg or ticagrelor 180 mg before surgery, and C13 breath test was performed after surgery.
* All patients were treated with dual- antiplatelet.
* The clinical data of the included subjects were complete.

Exclusion Criteria:

* Patients with previous liver and kidney disease, Cr greater than 150 μmol / L, AST or ALT increased more than 2 times the normal value of patients.
* Patient with history of cerebrovascular disease.
* Patients with active gastrointestinal bleeding disease due to cirrhosis or other reasons before PCI.
* Patients with abnormal coagulation.
* Diabetic patients, diagnostic criteria for anemia: 8th edition of internal medicine, adult males with Hb less than 120g / L or RBC less than 4 × 10^12 / L, adult women with Hb less than 105g / L or RBC than 3.5 × 10^12 / L.
* Patients with incomplete medical records;7.Patient with pregnant.
* Patients with malignant tumors

Ages: 24 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of acute myocardial infarction who need dual- antiplatelet after PCI.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
symptoms of upper gastrointestinal bleeding | 2019-12
  Number of participants with digestive discomfort, such as abdominal pain, nausea, belching, acid reflux, etc.
endoscopy examination of upper gastrointestinal bleeding | 2019-12
  Number of participants with spotted, linear or diffuse bleeding
the fecal examination of upper gastrointestinal bleeding | 2019-12
  Number of participants with melea, tar-like stool, hematemesis, fecal occult blood, etc.

CONTACTS AND LOCATIONS:
Overall Officials: DZhang D Z, Associate Professor, Principal Investigator — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No